CLINICAL TRIAL: NCT05043948
Title: Genome-wide Association Study of Development of Collateral Circulation for Patients With Coronary or Peripheral Artery Disease
Acronym: GWAScollateral
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jung-min Ahn (Other)
Responsible Party: Sponsor-Investigator, Jung-min Ahn, Assistant Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: GWAS_collateral
Record Dates: First submitted 2021-09-12; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Coronary Disease; Peripheral Arterial Disease; Collateral Circulation, Any Site
Keywords: Genome-wide association; Collateral circulation
MeSH Terms: conditions — Coronary Disease; Peripheral Arterial Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Coronary Artery Disease_collateral flow grade 2
  Interventions: Diagnostic Test: Blood samples
- Coronary Artery Disease_collateral flow grade 0
  Interventions: Diagnostic Test: Blood samples
- Peripheral Artery Disease_collateral flow grade 2
  Interventions: Diagnostic Test: Blood samples
- Peripheral Artery Disease_collateral flow grade 0
  Interventions: Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: Blood samples — for evaluation of the genome-wide association study

SUMMARY:
The purpose of this study is to evaluate the genome-wide association for the development of collateral circulation for patients with coronary or peripheral artery disease and to develop the molecular genetic treatment model based on genome-wide association data.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 20
* Chronic total occlusive lesion from the coronary or peripheral angiogram

Exclusion Criteria:

* Renal dysfunction
* Hepatic dysfunction
* Thrombocythemia or thrombocythemia
* Planned major surgery in 1 year
* History of gastrointestinal haemorrhage
* Malignant tumor

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic total coronary or peripheral occlusion
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-08-21 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between genome and collateral flow | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided